CLINICAL TRIAL: NCT06844357
Title: A Multi-center, Randomized, Controlled, Open-label Phase II/III Clinical Trial to Investigate Whether Transarterial Tirapazamine Injection Followed by Transarterial Embolization (TATE) is Superior to Traditional Transarterial Chemoembolization (TACE) in Patients With Intermediate-Stage Hepatocellular Carcinoma (HCC)
Brief Title: A Phase II/III Trial Comparing Transarterial Tirapazamine Embolization (TATE) With cTACE for Intermediate-stage Liver Cancer.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zhejiang Raygene Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RG001
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: HCC
MeSH Terms: interventions — Tirapazamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TATE (Experimental): Patients will receive a fixed dose of 35 mg tirapazamine via hepatic arterial injection, followed by embolization with iodized oil, gelatin sponge and contrast agent suspension.
  Interventions: Drug: tirapazamine; Procedure: Transarterial Embolization (TAE)
- TACE (Experimental): Patients will receive cTACE with a mixture of iodized oil （10mL）and epirubicin (50 mg ), followed by embolization with gelatin sponge and contrast agent suspension.
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: tirapazamine — Intra-arterial injection into the tumor feeding artery
  Arms: TATE
Procedure: Transarterial Embolization (TAE) — Lipiodol and Gelfoam used to embolize tumor vessels and induce tumor hypoxia
  Arms: TATE
Procedure: TACE — TACE with epirubicin
  Arms: TACE

SUMMARY:
This phase I/II clinical trial aims to determine the efficacy and safety of TATE compared to TACE in patients with intermediate-stage HCC. The results will provide valuable insights into the potential benefits of TATE as a novel treatment option for HCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary hepatocellular carcinoma according to AASLD criteria.
* No evidence of extrahepatic metastasis, regional lymph node involvement, or vascular tumor thrombus.
* Patients must be eligible for TAE or TACE treatment.
* ECOG ≤ 1.
* Child-Pugh score ≤ 7.
* Adequate bone marrow, liver, and kidney function is required.

Exclusion Criteria:

* History of liver transplantation.
* Previous radioemblization or radiotherapy for liver tumors.
* severe cardiovascular or renal diseases, active systemic infections.
* Clinically significant hypoxia (oxygen saturation < 92% without oxygen supplementation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 36 months
  Progression-free survival (PFS) assessed by the Independent Radiology Committee (IRC) using mRECIST criteria.

SECONDARY OUTCOMES:
Complete Response (CR) rate | 36 months
  Complete response rate (CR) assessed by IRC using mRECIST criteria
objective response rate (ORR) | 36 months
duration of complete response (DOCR) | 36 months
overall survival (OS) | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun Teng, M.D, Principal Investigator — Zhongda Hospital; Jiansong Ji, M.D, Principal Investigator — The Central Hospital of Lishui City
Locations (2):
- China (2):
  - Zhongda Hospital, Affiliated to Southeast University, Nanjing, Jiangsu
  - Lishui Central Hospital, Lishui, Zhejiang

IPD SHARING:
Plan to Share IPD: No
Privacy Protection for Participants